CLINICAL TRIAL: NCT06873555
Title: Phase Ib/IIa Multicenter, Open-Label Study to Evaluate the Efficacy, Safety, and Pharmacokinetic Profile of DC05F01 in Patients with Recurrent/Refractory Ovarian Cancer and Other Advanced Solid Tumors
Brief Title: A Study of DC05F01 in Chinese Patients with Recurrent/Refractory Ovarian Cancer and Other Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Heronova Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHRC-DC05F01-02
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumors; Ovarian Cancer; Small Cell Lung Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part A Cohort1 (Experimental): Patients with recurrent/refractory ovarian cancer will receive oral 2100 mg DC05F01 once daily, continuously, with a 4-week treatment cycle
  Interventions: Drug: DC05F01
- Part A Cohort2 (Experimental): Patients with limited-stage small cell lung cancer will receive oral 2100 mg DC05F01 once daily, continuously, with a 4-week treatment cycle
  Interventions: Drug: DC05F01
- Part A Cohort3 (Experimental): Patients with other advanced malignant solid tumors will receive oral 2100 mg DC05F01 once daily, continuously, with a 4-week treatment cycle
  Interventions: Drug: DC05F01
- Part B (Experimental): Patients with specific advanced malignant solid tumors will receive oral 2100 mg DC05F01 once daily, continuously, with a 4-week treatment cycle
  Interventions: Drug: DC05F01

INTERVENTIONS:
Drug: DC05F01 — DC05F01 capsule

SUMMARY:
This study is a multicenter, open-label, cohort expansion Phase Ib/IIa trial designed to evaluate the efficacy, safety, and pharmacokinetic (PK) profile of DC05F01 in patients with recurrent/refractory ovarian cancer and other advanced solid tumors.

DETAILED DESCRIPTION:
The study consists of two parts. Part A will expand the Phase I study based on safety, tolerability, pharmacokinetic characteristics, and preliminary efficacy data to select the recommended Phase II dose (RP2D, tentatively set at 2100 mg). The study plans to enroll 10 patients with recurrent/refractory ovarian cancer into Cohort 1, 10 patients with limited-stage small cell lung cancer who have not progressed after chemoradiotherapy into Cohort 2, and 20 patients with other advanced malignant solid tumors into Cohort 3. All patients will receive oral DC05F01 once daily, continuously, with a 4-week treatment cycle to assess the efficacy, safety, and pharmacokinetic profile of DC05F01.

Part B will be determined based on the efficacy and safety data from Part A, with the investigator and sponsor jointly deciding on the appropriate indications for further expansion. It plans to enroll 20 patients to further evaluate the efficacy and safety of DC05F01.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed the informed consent form, understanding the study and willing to follow and capable of completing all trial procedures.
2. Aged ≥18 years, regardless of gender.
3. Patients with locally advanced or metastatic disease, including:

   Cohort 1: Epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer with FIGO stage III-IV, previously treated with platinum-based therapy and experienced disease progression or recurrence during or within 6 months (184 calendar days) after the last platinum-based treatment.

   Cohort 2: Limited-stage small cell lung cancer patients, as staged by the Veterans Administration Lung Study Group (VALG), who are not surgical candidates and have not progressed during or after at least 4 cycles of platinum-based chemotherapy combined with concurrent or sequential radiotherapy, completed within 6 weeks before the first dose.

   Cohort 3: Other solid tumors that have failed standard treatment, have no standard treatment options, or for whom standard treatment is not applicable at present.
4. Cohort 1: Patients must have undergone initial or interval debulking surgery. Elevated CA125 alone without radiological or clinical evidence cannot be considered as disease progression or recurrence. Prior treatment may include bevacizumab and PARP inhibitors.

   Cohort 2: Chemotherapy regimens must include platinum agents and intravenous etoposide, followed by a radical radiotherapy regimen. Prophylactic cranial irradiation is allowed based on the investigator's judgment and local standard of care, completed within 6 weeks before the first dose.
5. According to RECIST 1.1 criteria, there must be at least one measurable lesion assessed by imaging (lesions within previously irradiated areas or treated with other local therapies are generally not considered measurable unless there is documented progression) (applicable to Cohort 1 and Cohort 3).
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
7. Expected survival time of ≥3 months.
8. No significant hematologic, hepatic, renal, coagulation, or cardiac function abnormalities. Laboratory test results during the screening period (no transfusions or hematopoietic growth factor support within 14 days before testing) must meet the following standards:

   Absolute Neutrophil Count (ANC) >1.5×10^9/L. Hemoglobin (HGB) ≥90 g/L. Platelets (PLT) >100×10^9/L. Total Bilirubin (TBIL) ≤1.5 mg/dL. Albumin (ALB): ≥3 g/dL. Aspartate Aminotransferase (AST)/Alanine Aminotransferase (ALT)/Alkaline Phosphatase (ALP)/Gamma-Glutamyl Transferase (GGT) ≤2.5 times the upper limit of normal (ULN). If liver metastases are present, AST/ALT/ALP < 5×ULN.

   Serum Creatinine (Scr) ≤1.5×ULN or Creatinine Clearance (CrCl) ≥60 mL/min. Prothrombin Time (PT)/Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN. Serum sodium, potassium, magnesium, calcium, and phosphate levels within normal range or deemed clinically insignificant by the investigator. Supplements to maintain normal electrolyte levels are permitted.
9. Male subjects and women of childbearing potential must agree to use effective contraception from the time of signing the informed consent form until 3 months after the last dose of the study drug. Women of childbearing potential must have a negative serum pregnancy test prior to the first dose of the study drug.

Exclusion Criteria:

1. Received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy, or other anti-tumor treatments within 4 weeks or 5 half-lives (whichever is shorter) before the first dose of the study drug, except for:

   Nitrosoureas or mitomycin C within 6 weeks before the first dose. Oral fluorouracil or small-molecule targeted drugs within 2 weeks or 5 half-lives (whichever is shorter) before the first dose.

   Anti-tumor traditional Chinese medicine within 2 weeks before the first dose.
2. Received any other investigational drug or treatment in another clinical trial within 4 weeks before the first dose.
3. Underwent major organ surgery (excluding biopsy) or significant trauma within 4 weeks before the first dose, or requires elective surgery during the trial period.
4. Used strong inhibitors or inducers of CYP3A4, CYP1A2, and/or CYP2D6 within 14 days or 5 half-lives (whichever is shorter) before the first dose.
5. Previous allogeneic hematopoietic stem cell or bone marrow transplantation, or previous solid organ transplantation, or current use of immunosuppressive drugs or anti-rejection medications.
6. Allergy to any active or inactive ingredient of the study drug.
7. Adverse effects from prior anti-tumor treatments have not resolved to ≤Grade 1 according to CTCAE v5.0 (except for toxicities deemed not to pose a safety risk by the investigator, such as alopecia, Grade 2 peripheral neuropathy, or stable hypothyroidism managed with hormone replacement).
8. Active hepatitis B (HBsAg positive with HBV-DNA > lower limit of detection at the study center); hepatitis C virus infection (HCV-RNA > lower limit of detection at the study center); positive HIV antibody test; positive Treponema pallidum antibody test.
9. Presence of brain metastases or leptomeningeal metastases during the screening period or previously.
10. Presence of uncontrolled third-space effusions (e.g., large pleural effusions and/or ascites) as judged by the investigator.
11. Severe cardiovascular diseases, including but not limited to:

    Serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, II-III degree atrioventricular block, etc.

    Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other Grade 3 or higher cardiovascular events within 6 months before the first dose.

    New York Heart Association (NYHA) functional class ≥II, or other high-risk structural heart diseases as judged by the investigator.

    Uncontrolled hypertension clinically (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg after treatment).

    Any factors increasing the risk of QTc prolongation or arrhythmias, such as heart failure, uncorrectable hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or use of any concomitant drugs known to prolong the QT interval.
12. Presence of active infections requiring systemic treatment within 4 weeks before the first dose.
13. Presence of gastrointestinal diseases affecting drug absorption, such as Crohn's disease, ulcerative colitis, or short bowel syndrome, in an acute exacerbation phase, which may affect the absorption, metabolism, or elimination of the study drug as judged by the investigator.
14. Presence of interstitial lung disease, pulmonary fibrosis, or drug-induced interstitial pneumonia, except for radiation-induced pneumonia.
15. Presence of other severe diseases, including liver disease, kidney disease, neurological/psychiatric disorders, endocrine system diseases, hematologic diseases, immune system diseases, etc., that may affect participation in the study as judged by the investigator.
16. Presence of other malignancies within the past 5 years, except for cured basal cell carcinoma of the skin, non-melanoma skin cancer, or in situ cervical cancer.
17. Known alcohol or drug dependence.
18. Presence of psychiatric disorders or poor compliance.
19. Pregnant or breastfeeding women.
20. Any other clinical or laboratory abnormalities or other reasons deemed by the investigator to make the subject unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 24 months
  Overall response rate (ORR) based on RECIST v1.1 as assessed by the investigator
Progression-free Survival (PFS) | Up to 24 months
  Progression-free survival (PFS) based on RECIST v1.1 as assessed by the investigator

SECONDARY OUTCOMES:
Number of Participants With Adverse Events | 24 months
  Incidence and severity of adverse events as assessed by CTCAE Version 5.0
PK profile of DC05F01 | From time zero up to 24 hours post-dose
  Peak Concentration (Cmax): The maximum plasma concentration of the drug.
PK profile of DC05F01 | From time zero up to 24 hours post-dose
  Area Under the Curve from Time Zero to the Last Measurable Concentration (AUC0-t): The area under the plasma concentration-time curve from time zero to the last measurable concentration.
PK profile of DC05F01 | From time zero up to 24 hours post-dose
  Area Under the Curve from Time Zero Extrapolated to Infinity (AUC0-∞): The area under the plasma concentration-time curve from time zero extrapolated to infinity.
PK profile of DC05F01 | From time zero up to 24 hours post-dose
  Time to Reach Peak Concentration (Tmax): The time at which the peak plasma concentration is reached.
PK profile of DC05F01 | From time zero up to 24 hours post-dose
  Elimination Half-Life (T1/2): The time required for the plasma concentration to decrease by half.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Fisrt Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Hunan Cancer Hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No